CLINICAL TRIAL: NCT01370226
Title: Optimizing Alcohol Brief Interventions in the ED: Computer vs. Clinician Delivery
Brief Title: Health Explorer - Optimizing Alcohol Brief Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Frederic C. Blow, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: AA018659; R01AA018659 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-09 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBI (Active Comparator): Computer delivered Brief Intervention
  Interventions: Behavioral: CBI
- TBI (Active Comparator): Therapist delivered Brief Intervention
  Interventions: Behavioral: TBI
- EUC (No Intervention): Enhanced Usual Care

INTERVENTIONS:
Behavioral: CBI — The multimedia, interactive Computer Brief Intervention (CBI) condition will be delivered using tablet computers. The content and format will be easily negotiated by participants. The 30-minute interventions are designed to address the primary target behavior of alcohol use, and will include a tailored review of participants' goals/values, feedback regarding their present alcohol use patterns and consequences (either actual experiences or potential based on risk behaviors), developing a discrepancy between their alcohol use and ability to meet goals and values through a decisional balance exercise, and formulation of a "change plan" tailored for each participant.
  Arms: CBI
Behavioral: TBI — Participants receive a 30-minute intervention session with a Master's-level clinician. The interventions are designed to address the primary target behavior of alcohol use, and will include a tailored review of participants' goals/values, feedback regarding their present alcohol use patterns and consequences (either actual experiences or potential based on risk behaviors), developing a discrepancy between their alcohol use and ability to meet goals and values through a decisional balance exercise, and formulation of a "change plan" tailored for each participant.
  Arms: TBI

SUMMARY:
The aims of the study are to develop and refine tailored motivational brief interventions that are parallel in structure but have varied delivery modalities (computer vs. therapist) for patients with at-risk or problematic alcohol use, and to conduct a randomized controlled trial comparing the efficacy of these BI approaches (CBI, TBI, control) on subsequent alcohol consumption and alcohol consequences, including alcohol-related injury, mental and physical-health functioning, and HIV risk behaviors at 3-, 6-, and 12-months post-ED visit.

DETAILED DESCRIPTION:
Although a high proportion of patients seen in Emergency Departments (EDs) have at-risk or problem alcohol use, few are screened and receive services such as brief interventions (BI) designed to help them cut-back or stop drinking. EDs do not routinely provide BIs, perhaps due to feasibility challenges such as training of staff, monitoring fidelity, and maintaining a system to ensure longer-term implementation. Alcohol BIs have been found to be efficacious and effective in a variety of health care settings. However, the evidence for their use in the ED has been mixed. There is a pressing need to develop efficacious strategies to screen and optimally deliver alcohol BIs in this fast-paced and widely-used setting. Existing clinician-delivered BI strategies need to be modified so that they can be standardized and administered with high fidelity and minimal demands on ED staff time and resources. Computer-delivered BIs are one method to address the challenges inherent in delivering interventions in this and other healthcare settings. The proposed study will use computerized screening via touch-screen computer tablets with audio to recruit inner-city ED patients screening positive for at-risk or problem alcohol use. Participants age 21-65 will be randomized to one of three conditions: 1) Computer-delivered brief intervention (CBI); 2) Therapist-delivered brief intervention (TBI); or 3) Enhanced usual care (EUC). All participants will receive written information regarding community resources; individuals who meet alcohol abuse/dependence criteria will also receive alcohol treatment referrals. Stratified random assignment [by gender; meeting criteria for an alcohol use disorder] will take place at baseline for all conditions. The rigorous examination of the efficacy of therapist- vs. computer-delivered BIs, including potential moderators and mediators, will address the key limitations raised by previous trials and will determine the optimal modality for wide implementation of brief alcohol interventions in this venue. Because the ED is such an important portal for entry into the medical care system, particularly for inner-city patients, the delivery of efficacious alcohol BIs that emphasize key motivational interviewing components and minimize staff resources could have a major public health impact.

ELIGIBILITY:
Inclusion Criteria:

* patients age 21-65 years presenting to the ED for medical care (except exclusions as noted below)
* ability to provide informed consent
* Additional criteria for intervention: past 3-month at-risk alcohol use

Exclusion Criteria:

* patients who do not understand English
* prisoners
* patients classified by medical staff as "Level 1 trauma" (e.g., unconscious, intubated on respirators, in need of immediate lifesaving procedures such as surgery)
* patients deemed unable to provide informed consent as stated above (e.g., intoxication, mental incompetence)
* patients treated in the ED for suicide attempts or sexual assault

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Alcohol use - number of drinking days | change over time (3, 6 and 12-months post baseline)
Alcohol use - number of drinks per day | change over time (3, 6 and 12-months post baseline)
Alcohol use - number of binge drinking days | change over time (3, 6 and 12-months post baseline)
Alcohol use | change over time (3, 6 and 12-months post baseline)
  Alcohol Use Disorders Identification Test (AUDIT-C)
Alcohol related consequences | change over time (3, 6 and 12-months post baseline)
  Consequences are measured using the modified Short Inventory of Problems (SIP).
Alcohol related consequences | change over time (3, 6 and 12-months post baseline)
  Consequences are measured using the Drinker Inventory of Consequences (DrInC)

SECONDARY OUTCOMES:
Consequences of Alcohol Use - injury | change over time (3, 6 and 12-months post baseline)
  Injury is measured using the Revised Injury Behavior Checklist (RIBC).
Consequences of Alcohol Use - health functioning | change over time (3, 6 and 12-months post baseline)
  Health functioning is measured using the Brief Symptom Index (BSI-18).
Consequences of Alcohol Use - health functioning - depression | change over time (3, 6 and 12-months post baseline)
  Depression is measured using the Patient Health Questionnaire (PHQ-9).
Consequences of Alcohol Use - HIV-risk behaviors | change over time (3, 6 and 12-months post baseline)
  HIV-risk behaviors measures include questions about condom use, number of sexual partners, sex under the influence.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System Emergency Department, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No